CLINICAL TRIAL: NCT01714973
Title: Phase I Randomized, Blinded Safety and Efficacy Trial of Amnion-derived Cellular Cytokine Solution (ACCS) Versus Saline Sprayed on the Breast of Women Undergoing Radiation Therapy for Breast Cancer After Surgical Removal of the Tumor
Brief Title: Study of ST266 Versus Saline in Treating Skin Irritation From Radiation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-02-12
Record Dates: First submitted 2012-10-16; First posted 2012-10-26 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Radiation-induced Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ST266 intact (Experimental): Ten (10) patients will be randomized before the first radiation treatment to receive ST266 (4ml) and saline placebo (4ml), one to the medial segment and the other to the lateral segment. The area of the breast will be divided into two, roughly equal parts, medial and lateral. The randomization scheme will be equal in each of two cohorts. The first cohort will receive ST266 and saline placebo applied to intact skin beginning immediately following the first radiation treatment, to continue immediately following each of ten (10) consecutive radiation treatments.
  Interventions: Biological: ST266
- ST266 inflamed (Experimental): Ten (10) patients will be randomized before the first radiation treatment to receive ST266 (4ml) and saline placebo (4ml), one to the medial segment and the other to the lateral segment. The area of the breast will be divided into two, roughly equal parts, medial and lateral. The randomization scheme will be equal in each of two cohorts. The second cohort will receive ST266 and saline placebo applied to inflamed skin (after inflammation is first noted) beginning immediately following the radiation treatment, to continue immediately following each of ten (10) consecutive radiation treatments.
  Interventions: Biological: ST266

INTERVENTIONS:
Biological: ST266 — Patients will receive ST266 spray, to half the breast and saline to the other half (blinded) after each of ten consecutive radiation therapy treatments. ST266 and saline will be sprayed onto the breast to deliver 0.01 ml/cm2.

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ST266 in treating radiation burns of the skin in patients undergoing treatments for breast cancer and to compare ST266 treated burns with those treated with saline placebo controls.

ELIGIBILITY:
Inclusion Criteria:

* A signed IRB - approved Informed Consent;
* Women 18 - 80 years of age;
* Biopsy-proven diagnosis of breast cancer with the tumor surgically removed.
* Whole breast radiation with or without ipsilateral axilla radiation therapy recommended by her radiation oncologist.
* If a woman is of child-bearing potential, she and her partner must use an effective form of birth control.
* Willing to participate in the clinical study and comply with the requirements of the trial.

Exclusion Criteria:

* Abnormal liver or kidney function studies being greater than 2x the upper limit of normal.
* Patients on hemodialysis
* Psychiatric condition or substance abuse which in the Investigator's opinion may pose a threat to patient compliance;
* History of non-compliance with treatment or clinical visit attendance.
* Participation in an investigational trial within 30 days of study entry.
* Women who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Significant Adverse Events (SAEs) | Start of therapy through six week follow-up visit

SECONDARY OUTCOMES:
Skin inflammation | start of therapy through six week follow-up visit
Quality of Life (QOL)scaled responses | start of therapy through one year follow-up
  Quality of Life (QOL) will be evaluated using a QOL Assessment (general to breast cancer patients receiving radiation therapy following tumor removal) and a QOL Supplement (specific to subjects receiving trial treatment). Both documents include subsets of questions, each with a different subscale. The assessments include both lifestyle QOL factors (sleep, activity, friends/family, general life enjoyment, etc.) and breast condition (pain, appearance, ect.). This secondary endpoint will focus on the QOL Supplement, comparing breast condition by treatment, noting changes in both the medial and lateral aspects breast including breast texture (thickening and hardness), pain, tenderness, shape, sensitivity, swelling, redness, itching, flaking skin, blistering and fluid leak. The patient will note, for each item, in which side of the breast they are experiencing the negative breast condition or if there is no difference.

OTHER OUTCOMES:
Cosmesis | 6 and 12 months post-treatment
  Cosmesis will be evaluated by photography and investigator assessment using the cosmesis form in National Surgical Adjuvant Breast and Bowel Project (NSABP) Protocol B-39, A Randomized Phase III Study of Conventional Whole Breast Irradiation Versus Partial Breast Irradiation for Women with Stage 0, I, or II Breast Cancer. The following factors will be evaluated in the skin: telangiectasia, atrophy, scarring, pigmentation, erythema, fat necrosis, and fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Trombetta, MD, Principal Investigator — West Penn Allegheny Health System; David L Steed, MD, Study Director — Noveome Biotherapeutics, formerly Stemnion
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No